CLINICAL TRIAL: NCT00326924
Title: Age of Red Blood Cells in Premature Infants Study (ARIPI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2004706-01H
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Results first posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Premature Birth
Keywords: Transfusion
MeSH Terms: conditions — Premature Birth | interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biological (Experimental): PRBCs that are less than 7 days old are considered 'fresh'.
  Interventions: Biological: Transfusion
- Standard PRBCs (Experimental): PRBCs 'stored' as per hospital policy.
  Interventions: Biological: Transfusion

INTERVENTIONS:
Biological: Transfusion — PRBC blood transfusions.
  Other Names: non applicable

SUMMARY:
To determine if the age of blood transfused to new borns in the NICU setting has an impact on their outcome.

ELIGIBILITY:
Inclusion Criteria:

* birthweight of less than 1250g
* admitted to participating NICU
* consent acquired from proxy for the patient

Exclusion Criteria:

* already received one or more transfusions
* requirement for an exchange transfusion
* will be receiving directed donations
* have rare blood types/difficult cross-match
* proxy has refused consent
* moribund on admission to NICU/expected to die
* mitigating child protection issues

Ages: 1 Minute to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 377 (Actual)
Dates: Start 2006-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Fergusson, PhD, Study Director — OHRI
Locations (1):
- Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Kekre N, Mallick R, Allan D, Tinmouth A, Tay J. The impact of prolonged storage of red blood cells on cancer survival. PLoS One. 2013 Jul 16;8(7):e68820. doi: 10.1371/journal.pone.0068820. Print 2013. PMID 23874777
- [Derived] Fergusson DA, Hebert P, Hogan DL, LeBel L, Rouvinez-Bouali N, Smyth JA, Sankaran K, Tinmouth A, Blajchman MA, Kovacs L, Lachance C, Lee S, Walker CR, Hutton B, Ducharme R, Balchin K, Ramsay T, Ford JC, Kakadekar A, Ramesh K, Shapiro S. Effect of fresh red blood cell transfusions on clinical outcomes in premature, very low-birth-weight infants: the ARIPI randomized trial. JAMA. 2012 Oct 10;308(14):1443-51. doi: 10.1001/2012.jama.11953. PMID 23045213
- [Derived] Fergusson D, Hutton B, Hogan DL, LeBel L, Blajchman MA, Ford JC, Hebert P, Kakadekar A, Kovacs L, Lee S, Sankaran K, Shapiro S, Smyth JA, Ramesh K, Bouali NR, Tinmouth A, Walker R. The age of red blood cells in premature infants (ARIPI) randomized controlled trial: study design. Transfus Med Rev. 2009 Jan;23(1):55-61. doi: 10.1016/j.tmrv.2008.09.005. PMID 19056034

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Biological | Standard PRBCs
Started | 188 | 189
Completed | 187 | 188
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biological | Standard PRBCs | Total
Number analyzed (Participants) | 188 | 189 | 377
Age, Continuous [Mean (Standard Deviation); unit: days] | 10.0 (9.7) | 9.9 (9.5) | 10 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 95 | 174
  Male | 109 | 94 | 203
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mothers' characteristics: White | 138 | 123 | 261
  Mothers' characteristics: Black | 17 | 24 | 41
  Mothers' characteristics: Latin American | 4 | 1 | 5
  Mothers' characteristics: Asian | 6 | 8 | 14
  Mothers' characteristics: Aboriginal | 10 | 20 | 30
  Mothers' characteristics: Filipino | 0 | 4 | 4
  Mothers' characteristics: Arab | 3 | 1 | 4
  Mothers' characteristics: Other or unknown | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  Canada | 188 | 189 | 377

OUTCOME MEASURES:

1. Primary Outcome: 1. Composite Outcome of Necrotizing Enterocolitis, Intraventricular Hemorrhage, Bronchopulmonary Dysplasia and Retinopathy of Prematurity at 30 and 90-days. 2. Mortality
Description: The primary outcome was a composite outcome composed of mortality and major neonatal morbidities associated with acute organ dysfunction or failure. In addition to death, the 4 major morbidities comprising the composite outcome were bronchopulmonary dysplasia, retinopathy of prematurity, necrotizing enterocolitis, and intraventricular hemorrhage.
Time Frame: 2 weeks, 4 weeks, 12 weeks, 90 days
Measure: Number; unit: participants
Arm/Group | Biological | Standard PRBCs
Number analyzed (Participants) | 188 | 189
participants | 99 | 100

2. Secondary Outcome: Clinically Suspected Infection and Culturally Confirmed Infections
Description: Infection was categorized as clinically suspected and positive cultures.
Time Frame: 90 days
Measure: Number; unit: number of participants
Arm/Group | Biological | Standard PRBCs
Number analyzed (Participants) | 188 | 189
number of participants | 146 | 146

3. Secondary Outcome: Length of Stay
Description: Length of Stay in neonatal intensive unit
Time Frame: until last participants left neonatal intensive care unit
Measure: Mean (Inter-Quartile Range); unit: number of days
Arm/Group | Biological | Standard PRBCs
Number analyzed (Participants) | 188 | 189
number of days | 84 [50 to 104] | 77 [50 to 104]

4. Secondary Outcome: Number of Participants Using Mechanical Ventilation.
Description: Number of Participants using Mechanical Ventilation
Time Frame: whether a mechanical ventilation was used at any time point during 90 days
Measure: Number; unit: participants
Arm/Group | Biological | Standard PRBCs
Number analyzed (Participants) | 188 | 189
participants | 151 | 153

ADVERSE EVENTS:
Arm/Group | Biological | Standard PRBCs
Serious Adverse Events (participants affected / at risk) | 0/188 | 1/189
Other Adverse Events (participants affected / at risk) | 0/188 | 0/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biological (N=188) | Standard PRBCs (N=189)
cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1) — One serious adverse event potentially related to transfusion was a diagnosis of cytomegalovirus infection in an infant randomized to the standard red cell group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes